CLINICAL TRIAL: NCT00826839
Title: A Randomized Controlled Trial of Treatment Protocols to Optimize Outcomes in Poor Responder In Vitro Fertilization (IVF) Patients: E2 Patch/Antagonist Protocol Versus OCP/Microdose Lupron Protocol
Brief Title: Oral Microdose Lupron Versus Luteal Estradiol Trial in Poor Responder In Vitro Fertilization (IVF) Patients
Acronym: OMLET
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0810010037
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Infertility
Keywords: In vitro fertilization; Poor responder patients; Randomized clinical trial; Estrogen patch; Gonadotropin-releasing hormone antagonist; Oral contraceptive pill; Microdose lupron
MeSH Terms: conditions — Infertility | interventions — Contraceptives, Oral; Oviol; Desogestrel; Leuprolide; Estradiol; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCP/MDL (Experimental): Oral contraceptive pills/microdose lupron
  Interventions: Drug: Oral contraceptive pill and microdose lupron
- E2/antagonist (Experimental): Estradiol patch/gonadotropin-releasing hormone antagonist
  Interventions: Drug: E2 patch/antagonist

INTERVENTIONS:
Drug: Oral contraceptive pill and microdose lupron — Desogestrel/ethinyl estradiol tablets, 0.15 mg/0.03 mg, one tablet by mouth daily for 14 days Leuprolide acetate 40 µg by subcutaneous injection twice a day during ovarian stimulation (approximately 14 days)
  Other Names: Ortho-Cept®; Desogen®; Reclipsen™; Apri®; Leuprorelin; Leuprorelin Acetate; Lupron
  Arms: OCP/MDL
Drug: E2 patch/antagonist — Estradiol transdermal system 0.1 mg/day (25 cm2 patch. Patch changed every other day x 3. Final patch left on for about 7 days. Total duration of therapy approximately 14 days.
  Gonadotropin-releasing hormone antagonist 0.25 mg subcutaneously every other day for 3 total doses.
  Other Names: Climara®; Ganirelix acetate injection®
  Arms: E2/antagonist

SUMMARY:
Hundreds of thousands of couples in the United States experience infertility each year. When initial measures do not help, some couples require a process called ovarian stimulation and in vitro fertilization (IVF). Usually, a woman produces at most one egg each month. Ovarian stimulation helps these women make more than one egg per month. However, this involves taking hormones that stimulate the ovary to produce many eggs at one time. The stimulatory hormones injected with a small needle. The eggs are removed from the ovary through a surgical procedure and then placed in a dish for fertilization by sperm to form embryos. The embryos are grown in the laboratory then replaced into the woman's uterus 3-5 days later.

The stimulation of the ovaries is important. Some patients undergo ovarian stimulation for IVF but do not respond to the treatment. This is a very difficult situation because even though several ovarian stimulation protocols have been used for poor responder patients, it is not clear which protocol works best. In fact, two of the most commonly used protocols have not been directly compared.

This study will randomize (like flipping a coin) couples with a history of low response who are going to start IVF treatment into two groups. In one group the female partner will use a protocol called "E2 patch/antagonist". These women will use an estrogen patch and injected antagonist for several days before starting injectable fertility medications. The other group will use a protocol called "OCP/microdose". This group of women will use oral contraceptive pills (OCPs) and small doses of lupron along with the other injectable fertility medications. We will then follow their progress to see how many eggs they produce and how many women get pregnant.

DETAILED DESCRIPTION:
Patients who have difficulty conceiving naturally often seek medical advice. These patients often undergo initial treatment with insemination using oral or injectable medications. However, if this fails to achieve a pregnancy, patients often undergo in vitro fertilization (IVF). IVF is a process which involves a protocol of injectable medications to stimulate the ovary to produce several eggs at once. These eggs are retrieved under ultrasound guidance and fertilized in the laboratory. After 3-5 days of growth in the laboratory, the appropriate number of embryos is then transferred back to the patient's uterus.

Sometimes, patients who go through ovarian stimulation and IVF do not respond well. These patients have low estrogen levels, few eggs retrieved, and fewer embryos to transfer back to the uterus. Overall, they have lower pregnancy rates than other patients. It is not clear which medication protocol would give them the highest chance of pregnancy. Two protocols, one called the "E2/antagonist" protocol and the other called the "OCP/microdose" protocol, are routinely used in poor responder patients. But, they have never been prospectively compared so it is not possible to say whether one approach is better.

In order to determine which medication protocol results in more pregnancies, we propose to randomize poor responder patients who are scheduled to undergo treatment with IVF to one of these two protocols. These two protocols are already standard care in IVF centers around the world. Following randomization, the clinical care of study participants will be the same as all other IVF patients. Specifically, the adjustment of medication, egg retrieval, and embryo transfer procedures will be identical to non-study patients undergoing IVF.

HYPOTHESIS We hypothesize that the poor responder patients undergoing ovarian stimulation for IVF with the E2/antagonist protocol will have a higher pregnancy rate than those in the OCP/microdose group.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for IVF who have a history of poor response as defined by one of the following:
* Cancellation of IVF due to inadequate follicular development
* Peak estradiol < 1000 pg/mL
* < 6 oocytes retrieved
* Age ≥18 years at the time of signing informed consent
* Availability of ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed)
* Willing and able to sign informed consent

Exclusion Criteria:

* Prior use of the E2/ganirelix or OCP/microdose protocol
* Less than 2 ovaries or any other ovarian abnormality
* Presence of uncorrected unilateral or bilateral hydrosalpinx
* Presence of any clinically relevant pathology affecting the uterine cavity or intramural fibroid ≥ 5cm
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, clinically significant ovarian cysts)
* Contraindications for the use of oral contraceptive pills (h/o thromboembolism, breast cancer, undiagnosed vaginal bleeding)
* Contraindications for the use of estrogen patches (h/o thromboembolism, breast cancer, undiagnosed vaginal bleeding)
* Abnormal karyotyping of the patient or her partner (if karyotyping is performed)
* Hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol
* Transfer of embryos to the patient not planned (i.e. gestational carrier use planned, embryos to be frozen)
* Unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 7 weeks gestation

SECONDARY OUTCOMES:
Cycle cancellation rate | Cycle completion
Peak estradiol level | Cycle completion
Ampules of gonadotropins required during ovarian stimulation | Cycle completion
Number of days of ovarian stimulation | Cycle completion
Number of oocytes retrieved | Cycle completion
Number of embryos transferred | Cycle completion
Number of embryos frozen | Cycle completion
Embryo grade | Cycle completion
Implantation rate | 7 weeks gestation
Miscarriage rate | 20 weeks gestation
Pregnancy outcome | Following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Zev Rosenwaks, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The Ronald O. Perlman and Claudia Cohen Center for Reproductive Medicine at Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: The Ronald O. Perlman and Claudia Cohen Center for Reproductive Medicine at Weill Cornell Medical College — http://www.ivf.org/